CLINICAL TRIAL: NCT03840720
Title: The Patient's Journey - Assessing the Time to Final Diagnosis in Patients With Neuroendocrine Tumors (NET) in Western Sweden
Brief Title: The Patient's Journey - the Time to Final Diagnosis in Patients With SiNET
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Andreas Hallqvist, Principal investigator, Vastra Gotaland Region
Other Study IDs: PR-1.0
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
"The patient's journey" is an interview based study assessing the patients' experience from the first symptoms to a final diagnosis focusing on patients with small intestinal neuroendocrine tumors.

DETAILED DESCRIPTION:
The project focus on patients with small intestinal neuroendocrine tumors (SiNET's) with an incidence of 1-2/100 000 yearly. The primary tumor(s) are often small and symptoms usually arise when the disease has become metastatic with hormonal symptoms and/or symptoms due to local growth. As the tumors grow slowly and the symptoms in many cases are rather diffuse and develops gradually over a long time period there is often a long delay from onset to a final diagnosis both depending on "patient's delay" and "doctor's delay" The aim of the current project is to map and analyze the patient's journey from the first appearance of symptoms to the time point of a final diagnosis and to try to identify factors contributing to a delayed process.

The method is interview based and the interviews will be analyzed through the Design Thinking Methodology

ELIGIBILITY:
Inclusion Criteria:

* Patients living in Western Sweden
* > 18 years of age
* Performance status 0-3
* Expected remaining survival of > 6 months
* Diagnosed with a small intestinal neuroendocrine tumor during 2016-2018

Exclusion Criteria:

* Not able to read and/or understand Swedish language
* Dementia/memory loss
* Performance status >3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in Western Sweden, > 18 years of age that has been diagnosed with a small intestinal neuroendocrine tumor during 2016-2018
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Initial symptoms | October 2019
  Mapping of patients initial symptoms and their time points through indepths interviews by design thinking methodology
Health care actions | October 2019
  Mapping of corresponding health care actions and their time points regarding the investigations of symptoms
Reasons for a delayed diagnosis | October 2019
  Mapping of herdles and delays in reaching a final diagnosis through design thinking methodology analysing the patients symptoms and the corresponding Health care actions

SECONDARY OUTCOMES:
Patients' efforts | October 2019
  Mapping of actions taken by the patient, trying to be diagnosed correctly, through indepths interviews by design thinking methodology

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Hallqvist, MD, PhD, Principal Investigator — Dept of Oncology, Sahlgrenska University Hospital, Gothenburg, Sweden
Locations (1):
- Dept of Oncology, Gothenburg, Sweden